CLINICAL TRIAL: NCT03736850
Title: A Phase I, Open Label, Multiple Dose, Dose Escalation and Expansion Study to Investigate the Safety, Tolerability, Pharmacokinetics and Antitumor Activities of the MEK Inhibitor CS3006 in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of CS3006 in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS3006-102
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-03

CONDITIONS: Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS3006 (Experimental)
  Interventions: Drug: CS3006

INTERVENTIONS:
Drug: CS3006 — In the dose escalation part, the dose levels will be escalated following a modified 3+3 dose escalation scheme.
  In the dose expansion part, participants will receive CS3006 at specified dose level(s).

SUMMARY:
This is a multicenter, open label, sequential-cohort, dose escalation & expansion phase I study to evaluate the clinical safety, tolerability, PK, and preliminary efficacy of CS3006 and to establish the Maximum Tolerated Dose (MTD）, if any, Recommended Phase II Doses (RP2Ds) and regimen of CS3006. The study is composed of two parts: Part 1 for dose escalation and Part 2 for dose expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for the trial.
2. Subjects must have a histologically or cytologically confirmed advanced or metastatic solid tumor(s) for which no effective standard therapy is available or tolerable.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy ≥ 12 weeks.
5. Able to swallow and retain oral medication.
6. Subject must have adequate organ function.
7. Use of effective contraception.

Exclusion Criteria:

1. Subjects receiving cancer therapy at the time of enrollment.
2. Has had prior chemotherapy, targeted therapy, immunotherapy or any other agents used as systemic treatment for cancer, within 14 days of the first dose of investigational product administration or who has not recovered from adverse events due to a previously administered agent.
3. Previous treatment with a MEK inhibitor.
4. Use of any investigational anti-cancer drug within 28 days before the first investigational product administration.
5. Current use of a prohibited medication.
6. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
7. Known brain metastasis or other CNS metastasis that is either symptomatic or untreated.
8. Primary malignancy of the central nervous system.
9. Evidence of severe or uncontrolled systemic diseases.
10. Subjects with clinically significant cardiovascular disease.
11. Human Immunodeficiency Virus (HIV) infection.
12. Subjects with active Hepatitis B or C infection.
13. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the investigational product or excipients.
14. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.
15. Unwillingness or inability to follow the procedures outlined in the protocol.

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From the day of first dose to 30 days after last dose of CS3006

CONTACTS AND LOCATIONS:
Locations (1):
- People's Liberation Army 307 Hospital, Beijing, Beijing Municipality, China